CLINICAL TRIAL: NCT02731378
Title: Combination With Intravenous Iron Supplementation or Doubling Erythropoietin Dose for Patients With Chemotherapy-induced Anaemia Inadequately Responsive to Initial Erythropoietin Treatment Alone
Brief Title: Erythropoietin and Iron Supplementation for Patients With Chemotherapy-induced Anaemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Chen Lin, Dr., Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016003
Record Dates: First submitted 2016-03-16; First posted 2016-04-07 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Chemotherapy-induced Anaemia
Keywords: erythropoietin; iron supplementation; inadequately responsive; chemotherapy-induced anaemia
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EPO plus sustained iron dextran (Experimental): Group 1, EPO treatment at the original dose plus IV iron dextran 200 mg every three weeks (Q3W) for 15 weeks
  Interventions: Drug: Erythropoietins (EPO); Drug: Sustained iron dextran supplementation
- EPO plus aggressive iron dextran (Experimental): Group 2, EPO treatment at the original dose plus IV iron dextran 100 mg, twice a week (BIW) for five weeks
  Interventions: Drug: Erythropoietins (EPO); Drug: Aggressive iron dextran supplementation
- Double EPO (Active Comparator): Group 3, the control group, doubling the EPO dose without preplanned iron supplementation
  Interventions: Drug: Erythropoietins (EPO)

INTERVENTIONS:
Drug: Erythropoietins (EPO) — A routine dose 10,000 IU of EPO, three times weekly by subcutaneous injections.
  Arms: EPO plus aggressive iron dextran; EPO plus sustained iron dextran
Drug: Aggressive iron dextran supplementation — Iron dextran 100 mg, BIW, through 90 minutes of IV infusion, for the first consecutive 5 weeks
  Arms: EPO plus aggressive iron dextran
Drug: Erythropoietins (EPO) — Doubling EPO dosage to 20,000 IU, three times weekly by subcutaneous injections with a maximum of 5 doses
  Arms: Double EPO
Drug: Sustained iron dextran supplementation — Iron dextran 200 mg, Q3W, through 90 minutes of IV infusion and a maximum of 5 doses
  Arms: EPO plus sustained iron dextran

SUMMARY:
A multicentre, randomized, open-label, parallel-group, active controlled non-inferiority study

DETAILED DESCRIPTION:
Chemotherapy-induced anaemia (CIA) is a significant health problem for patients with cancer undergoing chemotherapy, causing fatigue and reducing quality of life (QoL). Up to 75% of cancer patients undergoing chemotherapy and/or radiotherapy reportedly experience mild-to-moderate anaemia (defined by a haemoglobin level of 9 to 11 g/dL). In clinical trials, erythropoietins (EPOs) have been shown to increase haemoglobin levels and improve anaemia and QoL in cancer patients. However, recent meta-analyses have highlighted possible safety issues regarding EPO exposure. Preclinical studies have pointed towards the role of EPO in augmenting tumorigenesis, metastasis, risk of thrombosis, and drug resistance in certain tumor types (e.g., breast cancer), as it can activate important antiapoptotic pathways targeted by current antineoplastic therapies, thus counteracting their effects. Current guidelines in western countries and China recommend restricted usage of EPOs and reduction / prevention of blood transfusions in the treatment of cancer-induced anaemia.

However, the inadequate response to erythropoietic therapy has not been well-characterized through rigorous studies and hence remains poorly handled in routine clinical practice. A major cause for not responding to EPO treatment is likely functional iron deficiency (FID), which is defined as a failure to provide iron to the erythroblasts despite sufficient iron stores. Patients with FID require supplementation of usable iron to optimize response to erythropoietic therapy, which might not be accomplished with oral iron. In a recent prospective, open-label trial, patients receiving epoetin alfa for CIA who were treated with IV iron dextran had a significantly greater Hb response compared with those receiving oral iron. Meanwhile, in patients with CIA and no iron deficiency, IV iron supplementation significantly reduced treatment failures to darbepoetin without additional toxicity. However, whether that IV iron supplementation increases the risk of disease progression, incidence of thrombosis and heart failure as well as iron overload, is under careful investigation. Though the association between IV iron and serious AEs and mortality remains unclear, Zitt et al. found that the use of IV iron was associated with a 22% reduction in mortality. Therefore, investigators designed this multicentre, randomized trial to investigate EPOs in combination with IV iron with regard to an increase of Hb levels in patients who have inadequate responses to initial treatment with routine doses of EPOs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Had histologically, cytologically or clinically diagnosed malignant tumour and measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1;
* Undergoing adjuvant or palliative chemotherapy with an expected survival of at least 3 months;
* Inadequately responsive or unresponsive to routine dosages of EPO treatment. Inadequate responders or nonresponders are defined as those CIA patients with an increase of Hb < 1g/dL after 4 weeks of treatment with 10, 000 IU of EPO, three times weekly by subcutaneous injection).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2;
* Are compliant and can understand the research and sign an informed consent form.

Exclusion Criteria:

* History of thromboembolism in the previous twelve months;
* Family history of hemochromatosis;
* Anaemia diagnosed with myelodysplastic syndrome or hematologic diseases such as Mediterranean anaemia;
* Received EPO treatment in the prior three months;
* Received erythrocyte suspension transfusion in the prior two weeks;
* Women who are pregnant or lactating;
* Have a history of hypertension or mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-04 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Hb response rate | up to week 15
  A CIA patient would be defined as an Hb responder to study treatment if either Hb concentration of this patient is at least 12 g/dL or there is an increase in Hb levels of more than 2-g/dL compared to baseline level without blood transfusions initiated in the previous 28 days.

SECONDARY OUTCOMES:
Proportions of patients requiring therapeutic blood transfusions | Within 15 weeks
Time-to-progression (TTP) | Baseline, week 15, and then once per 3 months in the first year and once per 6 months thereafter up to 2 years
Volume of transfused blood | Within 15 weeks

OTHER OUTCOMES:
Adverse events (AEs) | Through study completion, up to 2 years
Quality of life - Linear Analogue Self-Assessment test | Baseline and week 3, 6, 9, 12 and 15
Quality of life - Functional Assessment of Cancer Therapy-Anaemia test | Baseline and week 3, 6, 9, 12 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Yong Gao, PhD, Principal Investigator — Shanghai East Hospital
Locations (6):
- China (6):
  - Shanghai East Hospital Home Branch, Shanghai, Shanghai Municipality
  - Shanghai East Hospital South Branch, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Lingang Branch, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, The Second Military Medical University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital Jian Branch, Jian, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen L, Jiang H, Gao W, Tu Y, Zhou Y, Li X, Zhu Z, Jiang Q, Zhan H, Yu J, Fu C, Gao Y. Combination with intravenous iron supplementation or doubling erythropoietin dose for patients with chemotherapy-induced anaemia inadequately responsive to initial erythropoietin treatment alone: study protocol for a randomised controlled trial. BMJ Open. 2016 Oct 7;6(10):e012231. doi: 10.1136/bmjopen-2016-012231. PMID 27855097